CLINICAL TRIAL: NCT06858410
Title: A Randomized, Open-label, Multicenter, Phase III Study of Lorlatinib Compared with Concurrent/ Sequential Chemoradiotherapy As Definitive Treatment in Patients with Locally Advanced, Unresectable Stage III ALK Positive Lung Adenocarcinoma
Brief Title: Lorlatinib Compared with Concurrent/ Sequential Chemoradiotherapy in Stage III ALK Positive Lung Adenocarcinoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Principal Investigator, Yi-Long Wu, Professor of Pulmonology, Guangdong Association of Clinical Trials
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTONG2403
Record Dates: First submitted 2025-02-19; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Neoadjuvant Non-Small Cell Lung Cancer
Keywords: ALK-positive; Stage III unresectable; Lung Adenocarcinoma; NSCLC
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — lorlatinib

STUDY DESIGN:
Intervention Model Description: A randomized, open-label, parallel study Lorlatinib compared with concurrent/ sequential chemoradiotherapy in locally advanced, unresectable Stage III ALK positive Lung Adenocarcinoma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- lorlatinib treatment (Active Comparator): In lorlatinib group, eligible patients will be registered to receive oral lorlatinib 100mg qd for 36 months during the treatment phase. Lorlatinib will be administered orally QD at approximately the same time of the day on a continuous daily dosing schedule, ie, without a break in dosing in the absence of drug-related toxicity
  Interventions: Drug: lorlatinib
- concurrent/sequential platinum-based chemoradiotherapy (Active Comparator): In concurrent/sequential platinum-based chemoradiotherapy group, the choice of chemotherapy and will be determined by the investigator prior to treatment allocation and the radiotherapy also according to the clinical therapy regimen decided by the investigator.
  Interventions: Other: concurrent/sequential platinum-based chemoradiotherapy

INTERVENTIONS:
Drug: lorlatinib — Eligible patients will be registered to receive oral lorlatinib 100mg qd for 36 months during the treatment phase.
  Arms: lorlatinib treatment
Other: concurrent/sequential platinum-based chemoradiotherapy — The choice of chemotherapy and will be determined by the investigator prior to treatment allocation and the radiotherapy also according to the clinical therapy regimen decided by the investigator.
  Arms: concurrent/sequential platinum-based chemoradiotherapy

SUMMARY:
The project is a Phase III, randomized, open-label, multicenter study in which approximately 36 patients with unresectable Stage III ALK positive Lung Adenocarcinoma will be randomized 1:1 to receive lorlatinib or concurrent/sequential platinum-based chemoradiotherapy

DETAILED DESCRIPTION:
Lung cancer is the most fatal malignancy in China, as estimated by National Cancer Center of China, accounting for 1,060,600 new cases, and 733,400 deaths in 2022. Non-small cell lung cancer (NSCLC) is the major pathological type of lung cancer, accounting for approximately 80%-85% of all lung cancer. Anaplastic lymphoma kinase (ALK) -positive NSCLC account for about 3%-7% of all non-small cell lung cancer.

30% of patients with NSCLC have reached stage III at the time of presentation, and most of these patients have lost the best opportunity for surgical treatment. Stage III NSCLC is a highly heterogeneous group of diseases that can be further divided into Stage IIIA, Stage IIIB, and Stage IIIC by TNM stage with 5-year survival rates of 36%, 26%, and 13%, respectively. Stage IIIA and a small proportion of stage IIIB NSCLC are classified as resectable, stage IIIC and the vast majority of stage IIIB are unresectable stage III NSCLC.

Prior guidelines recommended that patients with unresectable Stage III NSCLC with PS0-1 be treated with concurrent chemoradiotherapy, with sequential chemoradiotherapy as an option for intolerant patients. Following the advent of the era of immunotherapy, the PACIFIC study first confirmed that sequential durvalumab following simultaneous chemoradiotherapy as consolidation therapy significantly improved patient survival in unresectable Stage III NSCLC patients, redrafting the clinical treatment landscape for such patients. In addition, based on the GEMSTONE-301 study, the Chinese Society of Clinical Oncology (CSCO) guidelines recommend Sugemalimab as consolidation therapy after simultaneous or sequential chemoradiotherapy.

The results of chemoradiotherapy remain controversial for driver-positive unresectable stage III NSCLC. Stage III EGFR-positive NSCLC has been shown to significantly reduce median PFS after radiotherapy compared to wild-type (9.6 vs. 12.0 months; HR 2.0, 95% CI: 0.9-4.2, P=0.003) and no significant difference in OS (29.4 vs 23.4 months, P=0.21) 36-37. Also, the median OS for EGFR-mutated tumors was shown to be longer compared to wild-type, although the difference was not statistically significant. At the same time, the proportion of distant metastasis in driver-positive NSCLC is higher after simultaneous chemoradiotherapy than wild-type. For brain metastases, the cumulative incidence of brain metastases was 33% at 3 years and 44% at 5 years. These data suggest that PFS in driver positive patients is worse than in negative patients following simultaneous chemoradiotherapy with stage III NSCLC, mainly due to recurrent distant metastases, particularly brain metastases. In addition, the side effects of chemotherapy cannot be ignored. A meta-analysis of 1205 patients with locally advanced NSCLC in 6 clinical trials showed a significant benefit of concurrent chemoradiotherapy over sequential chemoradiotherapy overall survival, but the toxicity response also increased with time.

Tyrosine kinase inhibitors (TKIs) for ALK significantly improve tumor response and overall survival in patients with ALK-positive NASLS compared with empirical chemotherapy. And from the first generation ALK-TKI to the third generation ALK-TKI, the survival of patients with ALK-positive NSCLC lung cancer is increasing. Crizotinib was the first ALK inhibitor approved for the treatment of ALK-positive NSCLC. Subsequently, the emergence of more second-generation ALK TKI, including alectinib, brigatinib, ceritinib, and ensartinib, significantly prolonged median disease-free progression survival (mPFS) in patients with NSCLC and increased the intracranial response rate. However, ALK-resistance mutations (e.g., I1171N, L1196M, and G1202R) and intracranial metastases inevitably lead to the emergence of resistance, which is a major cause of death. The third-generation ALK-TKI lorlatinib CROWN study included the efficacy of treatment-naïve patients with ALK-positive advanced NSCLC compared to lorlatinib (n=149) and crizotinib (n=147). At follow-up 60.2 months, the median progression-free survival time (mPFS) remained NR (95% CI, 64.3-NR) in the lorlatinib arm and the mPFS was 9.1 months (95% CI, 7.4-10.9 months) in the crizotinib arm, with a hazard ratio of HR=0.19 (95% CI, 0.13-0.27). 5-year PFS was 60% (95% CI, 51 to 68) and 8% (95% CI, 3 to 14), respectively. Corresponding to the longest PFS ever reported with any single-agent molecular targeted treatment in advanced NSCLC and across all metastatic solid tumors and set a new benchmark for targeted therapies in cancer.

Based on the above background, there's a hypothesis that for ALK-positive Stage III unresectable Lung Adenocarcinoma, lorlatinib with high-potency inhibition, high CNS penetration, and broad-spectrum activity, may provide a superior survival benefit to these patients compared with chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Study Population: Patients with histologically or cytologically confirmed diagnosis of ALK-positive, lung adenocarcinoma who present with locally advanced, unresectable (Stage III) disease (according to Version 8 of the International Association for the Study of Lung Cancer [IASLC]).
* Tumor Requirements: At least 1 measurable target lesion per RECIST v. 1.1
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0-1. Life expectancy at least 12weeks at Day1.
* Age ≥18 years.
* Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Previously received any ALK-TKIs or any thoracic radiotherapy
* Active infection, including Bacteria, fungi or viruses
* Any evidence of severe or uncontrolled systemic diseases, which in the Investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardise compliance with the protocol
* Inadequate bone marrow reserve or organ function.

  1. Absolute neutrophil count <1.5*109/L
  2. Platelet count <90*109/L
  3. Hemoglobin <90 g/L (<9 g/dL) d Alanine aminotransferase > 3 times the upper limit of normal (ULN)

  e. Aspartate aminotransferase > 3 times the upper limit of normal (ULN) f. Total bilirubin > 1.5*ULN g. Creatinine >1.5*ULN or creatinine clearance <45 mL/min (calculated by Cockcroft-Gault formula)
* History of interstitial lung disease (ILD) or active ILD or pneumonia
* Pregnant female patients; breastfeeding female patients; fertile male patients and female patients of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 97 days, if male or 35 days if female, after the last dose of investigational product under lorlatinib.
* Participation in other studies involving investigational drug(s) within 2 weeks prior to study entry and/or during study participation.
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2030-03 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | up to 36 months from date of randomization until the date of first documented progression or date of death from any cause, whichever came first
  Progression Free Survival (PFS) is defined as the time from start of lorlatinib treatment to the date of disease progression as defined by RECIST v1.1 per investigator review or death due to any cause, whichever occurred first

CONTACTS AND LOCATIONS:
Overall Officials: E E Ke, M.D., Study Chair — Guangdong Provincial People's Hospital

IPD SHARING:
Plan to Share IPD: No